CLINICAL TRIAL: NCT04382716
Title: Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS): Clinical Characterization and Prospective Course
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: University_of_Minnesota
Record Dates: First submitted 2020-04-23; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: PANS; PANDAS
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PANS participants
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; observation only

SUMMARY:
This study is a brief (3 month) longitudinal study following children between the ages of 4-16 years old who have been diagnosed with Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS). Parents and children (who are at a 2nd grade reading level) will complete questionnaires online or in person weekly for 3 months. Additionally, parents will track their child's symptoms 3 times/week using a mobile application for 3 months. The investigators are hoping to begin to characterize the longitudinal trajectory of neuropsychiatric symptoms in children with PANS. Additionally, the study will seek to identify baseline demographic and clinical characteristics (e.g., gender, recent onset versus chronic course, GAS versus other triggers) that predict severity of baseline neuropsychiatric symptoms and predict change in symptoms over time.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking boys and girls ages 4-16 years
* Abrupt onset of OCD or severely restricted food intake
* At least 2 equally abrupt-onset concurrent neuropsychiatric symptoms from the following 7 categories: anxiety, emotional lability/depression, irritability/aggression/severely oppositional behaviors, behavioral/developmental regression, deterioration in school performance, sensory or motor abnormalities (e.g. tics), somatic symptoms (e.g., urinary, sleep)
* Neuropsychiatric symptoms are not better explained by a known neurological or medical disorder.

Exclusion Criteria:

- Too unstable psychiatrically or medically to participate safely in the protocol, per clinical judgment of the Principal Investigator or Co-Investigator

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with an established or suspected diagnosis of PANS/PANDAS.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale Compliance | Week 12
  Investigators will report overall compliance rates (percentage of completed questionnaires) for the Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale.
Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale Agreement | Week 12
  Investigators will also report agreement between parent and child Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale total scores across the study. Agreement will be reported using correlations.
Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale Predictors | Week 12
  Investigators will report items from the baseline Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) Symptom Rating Scale that predict symptom severity across the study using a regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harris EC, Conelea CA, Shyne MT, Bernstein GA. Predictors and Prospective Course of PANS: A Pilot Study Using Electronic Platforms for Data Collection. J Child Adolesc Psychopharmacol. 2021 Mar;31(2):102-108. doi: 10.1089/cap.2020.0124. Epub 2020 Dec 31. PMID 33395354